CLINICAL TRIAL: NCT02420860
Title: Phase II Study of the Combination of Elotuzumab With Lenalidomide as Maintenance Therapy Post Autologous Stem Cell Transplant in Patients With Multiple Myeloma
Brief Title: Elotuzumab and Lenalidomide After Stem Cell Transplant in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0729; NCI-2015-00762 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0729 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic Cell Transplantation Recipient; Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (elotuzumab, lenalidomide) (Experimental): Patients receive elotuzumab IV over 2-4 hours on days 1, 8, 15, and 21 of courses 1-2 and on day 1 of each subsequent course. Patients also receive lenalidomide PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Elotuzumab; Drug: Lenalidomide; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Elotuzumab — Given IV
  Other Names: BMS-901608; Empliciti; HuLuc-63; HuLuc63; PDL-063; PDL063
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well elotuzumab works when given with lenalidomide as maintenance therapy after transplant in patients with newly diagnosed multiple myeloma who underwent transplant using their own stem cells (autologous transplant). Maintenance therapy is treatment that is given to help keep cancer from coming back after it has disappeared following the initial treatment. Immunotherapy with monoclonal antibodies, such as elotuzumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Biological therapies, such as lenalidomide, may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Adding elotuzumab to standard maintenance therapy with lenalidomide may work better in treating patients with multiple myeloma who have undergone transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish activity of elotuzumab and lenalidomide in the maintenance setting post autologous stem cell transplant (ASCT) in myeloma patients.

II. Progression free survival (PFS).

SECONDARY OBJECTIVES:

I. Progression free survival 2. II. Overall survival. III. Determine incidence of secondary primary malignancy. IV. Evaluate the best response rate (stringent complete response [sCR]/very good partial response [VGPR]/partial response [PR]) based on International Myeloma Working Group (IMWG) criteria.

V. Evaluate time to progression. VI. Evaluate time to next therapy. VII. Evaluate the tolerability and toxicity. VIII. Perform MD Anderson Symptom Inventory (MDASI)-Myeloma symptom evaluation.

OUTLINE:

Patients receive elotuzumab intravenously (IV) over 2-4 hours on days 1, 8, 15, and 21 of courses 1-2 and on day 1 of each subsequent course. Patients also receive lenalidomide orally (PO) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have undergone autologous stem cell transplantation, within 18 months of initiation of induction therapy for newly diagnosed myeloma
* Time to initiation of maintenance therapy: patients may start maintenance therapy as early as 60 days post-transplant and up to 210 days post-transplant; as long as they meet the following criteria:
* Platelet count >= 100,000/mm^3
* Neutrophil count >= 1000/mm^3 (no growth factors within 5 days)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Creatinine < 2.5 mg/dl
* Recovered (i.e., =< grade 1 toxicity) from the reversible effects of autologous stem cell transplant
* Patients whose primary therapy was changed due to suboptimal response or toxicity will be eligible, however no more than 2 regimens will be allowed prior to ASCT
* Patients must have an Eastern Cooperative Oncology Group (ECOG) status of 0 to 2
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female patients who: are postmenopausal for at least 24 months before the screening visit, OR; are surgically sterile, OR; if they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, 28 days prior to starting study drug, during study treatment and for 28 days after the last dose of study treatment, OR agree to completely abstain from heterosexual intercourse; male patients, even if surgically sterilized (i.e., status post vasectomy), who: agree to practice effective barrier contraception during the entire study treatment period and through 28 days after the last dose of study treatment, OR; agree to completely abstain from heterosexual intercourse

Exclusion Criteria:

* Major surgery within 14 days before the first dose of study drug
* Radiotherapy within 14 days before enrollment
* Known active central nervous system involvement
* Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment
* Female subject is pregnant or lactating
* Known active hepatitis B virus hepatitis, or known active hepatitis C virus
* Infection requiring systemic IV antibiotic therapy within 7 days before cycle 1 day 1 of therapy
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations
* Failure to have fully recovered (i.e., =< grade 1 toxicity) from the effects of prior chemotherapy regardless of the interval since last treatment
* Co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | The time from autologous stem cell transplantation to the time of clinical progression, death, whichever occurs first or the time of last contact, assessed up to 48 months
  Will be estimated using the Kaplan-Meier method. The log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model may be used to include multiple covariates in the time-to-event analysis.

SECONDARY OUTCOMES:
Response rate | Up to 48 months
  Estimated along with 95% confidence intervals.
Incidence of new primary malignancy | Up to 48 months
  Estimated along with 95% confidence intervals.
Overall survival | Up to 48 months
  Will be estimated using the Kaplan-Meier method. The log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model may be used to include multiple covariates in the time-to-event analysis.
Incidence of toxicity | Up to 48 months
  Toxicity data will be summarized by frequency tables. Per-treated analysis will be used to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received. The intensity (severity) of adverse events will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Sheeba Thomas, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org